CLINICAL TRIAL: NCT01813318
Title: Double-Blind Placebo-Controlled Study of Acamprosate in Autism
Brief Title: Study of Acamprosate in Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CIN001-Acamprosate in Autism
Record Dates: First submitted 2013-01-30; First posted 2013-03-18 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2020-03

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo/sugar pill (Placebo Comparator): Placebo will be dosed similar to acamprosate, in terms of dosage form, frequency and duration.
  Interventions: Drug: Placebo
- Acamprosate (Active Comparator): Acamprosate: The maximum dose of acamprosate to be used in this study is 1998 mg per day for those subjects weighing greater than 50kg and 1332 mg per day for those less weighing less than 50kg.
  Other Name: Campral
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate — The maximum dose of acamprosate to be used in this study is 1998 mg per day for those subjects weighing greater than 50kg and 1332 mg per day for those less weighing less than 50kg.
  Other Names: Campral
  Arms: Acamprosate
Drug: Placebo — Subjects receiving placebo will be dosed similarly to the acamprosate group.
  Arms: Placebo/sugar pill

SUMMARY:
Recent pharmacotherapy research in autism spectrum disorders (ASD) has successfully focused on treatment of co-occurring symptoms, including inattention, hyperactivity, and irritability that commonly occur in persons with ASD. Despite over two decades of significant pharmacotherapy research, to date no medication has been shown in controlled trials to enhance the core social deficits of ASD. Based upon findings describing the neurobiology of ASD combined with our preliminary results, we believe the novel drug acamprosate will show evidence of reducing social skills deficits associated with ASD.

DETAILED DESCRIPTION:
Each subject with ASD will receive 10 weeks of blinded treatment with acamprosate or matching placebo. After completion of the double-blind phase, all subjects will have an opportunity to receive acamprosate as part of the study procedures for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 5-17 year-old outpatients
* Diagnosis of ASD
* General good health (determined by exam, history, and laboratory work up)
* Use of up to two concomitant psychotropic drugs (stable dosing for >60 days) not impacting glutamate or gamma-aminobutyric acid A (GABA) neurotransmission is allowed
* Stable seizure disorder (no seizures in 6 months; on same anti-convulsant dose for >60 days)
* Clinical Global Impression Scale Severity score (CGI-S) of 4 (Moderately III)
* Score of 13 on the Social Withdrawal subscale of the Aberrant Behavior Checklist (ABC-SW) at screen and baseline

Exclusion Criteria:

* Potential subjects with a creatinine clearance < 50 mL/min or evidence of a previous trial of acamprosate will be excluded

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 10 on the Social WIthdrawal subscale of ABC | Week 10
  The subscales of the ABC including the Social Withdrawal subscale have proven to be reliable measure of symptoms and behaviors associated with ASD. Specifically, the ABC-SW has been validated as a measure of social impairment that differentiates the social behavior of persons with ASD from those developmental delay without a comorbid ASD diagnosis.
Change Clinical Global Impression- Improvement | Week 10
  The CGI-I is a 7-point scale designed to measure symptomatic change at a specific time as compared to baseline. The CGI-I will be focused on the target symptoms of social impairment.

SECONDARY OUTCOMES:
Change in ABC subscales: Irritability, Stereotypy, Hyperactivity, and Inappropriate Speech from baseline to week 10 | Week 10
  The subscales of the ABC including the Social Withdrawal subscale have proven to be reliable measure of symptoms and behaviors associated with ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Erickson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States